CLINICAL TRIAL: NCT07217678
Title: Biomarkers of Ocular Surface Damage in the Setting of Topical Ocular Hypotensive Medication Use
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Swarup Swaminathan, Associate Professor of Ophthalmology, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240111
Record Dates: First submitted 2025-10-14; First posted 2025-10-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Glaucoma; Open-Angle Glaucoma; Ocular Hypertension; Glaucoma Suspect
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Durysta (Experimental): Participants will receive a one-time intracameral administration of Durysta - bimatoprost 10mcg
  Interventions: Drug: Durysta, Bimatoprost Intracameral Implant 10 µg

INTERVENTIONS:
Drug: Durysta, Bimatoprost Intracameral Implant 10 µg — Participants in this arm will receive a one-time injection of Durysta (intracameral bimatoprost 10mcg). Participants will be followed by a total of 3 months.

SUMMARY:
The objective of this study is to evaluate whether reduction in topical medication with the injection of a sustained release capsule (Durysta) leads to a reduction in ocular surface inflammation, indicated by levels of caspase-1, an inflammatory biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Eye with open-angle glaucoma or suspected of open-angle glaucoma
* Pseudophakic in eye of interest with Shafer grading ≥3
* ≤ 3 daily applications of topical glaucoma medications for ≥6 months (of which one is a nightly preserved PGA)
* Good adherence to medication regimen - screening questions to be asked of potential subject:
* In the last month, what percentage of the time would you estimate missing the application of drops? (Must be ≤20%)
* When was the last administration? (Last dose must have been within last 24 hours)
* Presence of punctate epithelial erosions in the cornea (NEI scale > 3)

Exclusion Criteria:

* Retinal disease (e.g., wet age-related macular degeneration, proliferative diabetic retinopathy, central retinal vein occlusion)
* Use of topical or systemic immunosuppressor or immunomodulator drug (e.g., steroids, cyclosporine, lifitegrast, or antihistamines)
* Use of preservative-free hypotensive medications
* Any clinical contraindications to receiving intracameral bimatoprost implantation
* History of recurrent conjunctivitis (e.g., allergic or atopic conjunctivitis)
* History of partial or full corneal transplant
* History of ophthalmic surgery (intraocular or tarsus-involving oculoplastic procedures) within last 6 months
* History of subconjunctival glaucoma surgery (i.e., trabeculectomy, aqueous shunt, Xen implant) within last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Caspase-1 mRNA Expression Following Durysta Injection | Baseline, post-injection 1 month, post-injection 3 months
  The primary outcome is evaluating whether the level of caspase-1 from the ocular surface changes after the Durysta injection when the number of topical medications is reduced. Higher values indicate more inflammation, while lower values indicate less information and a more stable ocular surface. The Caspase-1 level will be measured using RT-PCR.

SECONDARY OUTCOMES:
Change in Corneal Sensitivity Following Durysta Injection | Baseline, post-injection 1 month, post-injection 3 months
  Change in corneal tactile sensitivity from measured using a non-contact esthesiometer (in sensitivity units). Greater sensitivity values indicate less ocular surface dysfunction; lower values reflect reduced sensitivity and potential surface.
Change in Ocular Pain Symptoms via Visual Analog Scale (VAS) | Baseline, post-injection 1 month, post-injection 3 months
  Change in patient-reported ocular pain symptoms from post-Durysta injection, assessed using a Visual Analog Scale (VAS). VAS scores range from 1 to 10, where higher scores indicate more severe pain and lower scores reflect minimal discomfort.
Change in Corneal Staining Score Using the National Eye Institute (NEI) Grading System | Baseline, post-injection 1 month, post-injection 3 months
  Change in corneal staining score post-Durysta injection, assessed using the National Eye Institute (NEI) grading system. This system evaluates five corneal regions-central, temporal, superior, nasal, and inferior-with each region scored from 0 to 3 based on fluorescein staining intensity. The total score ranges from 0 (no staining) to 15 (diffuse staining across all regions). Lower scores indicate improved ocular surface integrity and reduced epithelial damage; higher scores reflect more extensive surface compromise.

CONTACTS AND LOCATIONS:
Overall Officials: Swarup S Swaminathan, MD, Principal Investigator — University of Miami
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No